CLINICAL TRIAL: NCT05598450
Title: rTMS for Auditory Hallucinations Guided by Magnetoencephalography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NDYX20220601
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2023-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation; Magnetoencephalography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- schizophrenia patients with auditory hallucinations (Experimental): For schizophrenia patients with auditory hallucinations, rTMS+MEG for implementation intervention
  Interventions: Device: rTMS and MEG for auditory hallucinations via self controlled clinical trials

INTERVENTIONS:
Device: rTMS and MEG for auditory hallucinations via self controlled clinical trials — a 4 weeks, weekly 345（23min*3times*5day） minutes, 1Hz, 100%RMT-rTMS protocol
  Detail precedure:
  Before intervention, each patient was scheduled to collect three magnetoencephalogram data sessions. Apply MEG technology to calculate possible locations and determine three intervention targets. Pseudo stimulation in the first week, 5-day intervention, 3 targets per day, each target for 23 minutes, with a 30 minute interval between each target. Evaluate the scale after the first week of pseudo stimulation. Week 2-4 real stimulation, intervention 5 days a week, 3 targets per day, each target for 23 minutes, with a 30 minute interval between each target. After the end of the fourth week, evaluate the scale. And follow-up evaluations will be conducted on the 7th, 14th, 30th, 60th, and 90th days after the intervention.

SUMMARY:
rTMS and MEG for auditory hallucinations via self controlled clinical trials. Repetitive transcranial magnetic stimulation (rTMS) can increase or decrease cortical excitability in patients with psychosis (such as schizophrenia). Here, we conducted an open clinical trial on 60 schizophrenics with auditory hallucinations. We searched for targets through magnetoencephalography and then intervened to prove that rTMS guided by magnetoencephalography is effective for auditory hallucinations.

DETAILED DESCRIPTION:
Before intervention, each patient was scheduled to collect three magnetoencephalogram data sessions. Apply MEG technology to calculate possible locations and determine three intervention targets. Pseudo stimulation in the first week, 5-day intervention, 3 targets per day, each target for 23 minutes, with a 30 minute interval between each target. Evaluate the scale after the first week of pseudo stimulation. Week 2-4 real stimulation, intervention 5 days a week, 3 targets per day, each target for 23 minutes, with a 30 minute interval between each target. After the end of the fourth week, evaluate the scale. And follow-up evaluations will be conducted on the 7th, 14th, 30th, 60th, and 90th days after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia with auditory hallucinations was diagnosed by DSM-IV, AHRS >12, Take sufficient antipsychotics for at least 1 month.

Exclusion Criteria:

* current pregnancy, major medical illness affecting the central nervous system, significant neurologic disorders, intake of drugs including supplements like essential fatty acids that influence prostaglandins or niacin skin flush flash pathway metabolism, a history of suicide risk, or alcohol or drug abuse.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Reduction rate of AHRS scale | One month
  Reduction rate of AHRS scale (the minimum is 0, maximum value is 47, and higher scores mean a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Yegang Hu, Doctor, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cash RFH, Weigand A, Zalesky A, Siddiqi SH, Downar J, Fitzgerald PB, Fox MD. Using Brain Imaging to Improve Spatial Targeting of Transcranial Magnetic Stimulation for Depression. Biol Psychiatry. 2021 Nov 15;90(10):689-700. doi: 10.1016/j.biopsych.2020.05.033. Epub 2020 Jun 7. PMID 32800379
- [Result] Lynch CJ, Elbau IG, Ng TH, Wolk D, Zhu S, Ayaz A, Power JD, Zebley B, Gunning FM, Liston C. Automated optimization of TMS coil placement for personalized functional network engagement. Neuron. 2022 Oct 19;110(20):3263-3277.e4. doi: 10.1016/j.neuron.2022.08.012. Epub 2022 Sep 15. PMID 36113473